CLINICAL TRIAL: NCT00829049
Title: Safety and Efficacy of Tazarotene Cream 0.1% Compared With Adapalene Gel 0.3% in the Treatment of Moderate to Severe Facial Acne Vulgaris
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study enrollment was terminated due to company decision before the target enrollment of 220 patients was reached.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-TAZ0702
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tazarotene Cream 0.1% (Active Comparator): 1 pea-size amount, QD x 16 weeks
  Interventions: Drug: Tazarotene Cream 0.1%
- Adapalene Gel 0.3% (Active Comparator): 1 pea-size amount, QD x 16 weeks
  Interventions: Drug: Adapalene

INTERVENTIONS:
Drug: Tazarotene Cream 0.1% — 1 pea-size amount, QD x 16 weeks
  Other Names: TAZORAC® Cream 0.1%
  Arms: Tazarotene Cream 0.1%
Drug: Adapalene — 1 pea-size amount, QD x 16 weeks
  Other Names: Differin® Gel 0.3%
  Arms: Adapalene Gel 0.3%

SUMMARY:
Comparison of the safety and efficacy of Tazarotene Cream 0.1% compared with Adapalene Gel 0.3% in treating moderate to severe facial acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Facial acne vulgaris characterized by the following: 25-100 facial inflammatory lesions (papules plus pustules); and 40 or more non-inflammatory lesions (open/closed comedones)); stable disease, non-rapidly regressing facial acne vulgaris; and, 3 or less facial nodules and/or cysts (diameter of 1cm or greater).
* Female subjects of childbearing potential must have a negative urine pregnancy test at baseline and practice reliable method of contraception throughout the study.

Exclusion Criteria:

* Non-compliance with washout period
* Skin disease/disorder that might interfere with diagnosis or evaluation of acne vulgaris
* Allergy or sensitivity to any component of the test medications
* Cosmetic or surgical procedure complementary to the treatment of facial acne within 14 days of the baseline visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Fremont, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Started | 77 | 88
Completed | 60 | 68
Not Completed | 17 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3% | Total
Number analyzed (Participants) | 77 | 88 | 165
Age Continuous [Mean (Full Range); unit: years] | 20.9 (7.7) [12.6 to 45.7] | 20.8 (7.6) [12.6 to 51.4] | 20.9 (7.6) [12.6 to 51.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 56 | 104
  Male | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change From Baseline in the Non-Inflammatory Lesion Counts (Open and Closed Comedones) at Week 12
Description: Median percent change from baseline in the non-inflammatory lesion counts (open and closed comedones) at Week 12. Comedones are small bumps on the skin (lesions) caused by acne and found at the opening of a skin pore. Open comedones (also known as blackheads) have a microscopic opening to the skin surface, while closed comedones (also known as whiteheads or pimples) lack the opening to the skin. A negative number change from baseline indicates a reduction in lesion counts(improvement).
Time Frame: Baseline, Week 12
Population: Intent to Treat population included all randomized patients. The number of patients that were analyzed reflects the actual number of patients for which data were available for this outcome measure.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Number analyzed (Participants) | 62 | 73
Percent Change | -68.14 [-96.23 to -2.99] | -60.00 [-100.00 to 42.86]

2. Secondary Outcome: Percentage of Patients With >= 1 Grade Improvement in the Investigator Global Assessment at Week 16
Description: Percentage of patients with >= 1 grade improvement (decrease in score) in the Investigator Global Assessment (IGA) at Week 16. The IGA is a 5-point scale used by the investigator to assess overall acne severity, where 0 equals clear skin (no evidence of acne) and 4 equals severe acne.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Number analyzed (Participants) | 61 | 72
Percentage of patients | 77.0 | 66.7

3. Secondary Outcome: Percentage of Patients With >= 2 Grade Improvement in the Overall Disease Severity Score at Week 12
Description: Percentage of patients with >= 2 grade improvement (decrease in score) in the overall disease severity score at Week 12. The overall disease severity score was evaluated by the investigator using a 7-point scale to rate the overall acne severity (lesions, inflammation, facial redness, and skin condition), where 0=no acne lesions and 6=most severe acne.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Number analyzed (Participants) | 61 | 73
Percentage of patients | 50.8 | 32.9

4. Secondary Outcome: Median Percent Change From Baseline in Inflammatory Lesion Counts (Papules/Pustules, Nodules) at Week 16
Description: Median percent change from baseline in inflammatory lesion counts (papules/pustules, nodules) at Week 16. Papules and nodules are round, solid elevations of the skin with no visible fluid; papules are smaller (less than 5 to 10 millimeters in width and depth) and nodules are larger (greater than 5 to 10 millimeters in width and depth). Pustules are small elevations of the skin containing cloudy material. A negative number change from baseline indicates a reduction in lesion counts (improvement).
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Number analyzed (Participants) | 61 | 72
Percent Change | -67.86 [-100.0 to 32.00] | -55.56 [-100.0 to 38.46]

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs an AEs and is the total number of patients that were randomized AND treated.
Arm/Group | Tazarotene Cream 0.1% | Adapalene Gel 0.3%
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/85
Other Adverse Events (participants affected / at risk) | 10/72 | 9/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tazarotene Cream 0.1% (N=72) | Adapalene Gel 0.3% (N=85)
Cold Symptoms (Infections and infestations) | 6 | 5
Burning (General disorders) | 4 | 4

LIMITATIONS AND CAVEATS:
Study enrollment was terminated due to company decision before the target enrollment of 220 patients was reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo